CLINICAL TRIAL: NCT06141395
Title: Development Of A Non-Interventional Diagnostic Ngs-Based Assay Of Blood Samples Of Sepsis Patients For Rapid Bacterial Identification Based On Next Generation Sequencing.
Brief Title: NGS-Based Assay of Blood Samples of Sepsis Patients for Rapid Bacterial Identification
Acronym: BIOARTE
Status: Completed | Type: Observational
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Collaborators: The BioArte (Unknown)
Responsible Party: Sponsor
Other Study IDs: BIOARTE
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-12

CONDITIONS: Pneumonia; Acute Pyelonephritis; Bacteremia; Biliary Tract Infection
Keywords: Bacterial Infection; Antimicrobial susceptibility testing; Next generation sequencing; Blood culture; Time to pathogen identification
MeSH Terms: conditions — Pneumonia; Bacteremia; Cholangitis; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an infection: Patients with high suspicion of infection with at least one sign of the quick Sequential Organ Failure Assessment (qSOFA) score
  Interventions: Diagnostic Test: NGS-based assay for bacterial identification

INTERVENTIONS:
Diagnostic Test: NGS-based assay for bacterial identification — A total volume of 26ml of whole blood will be sampled from each enrolled patient for three consecutive days. This will be used for Standard-of-Care (SoC) culture and Next Generation Sequencing (NGS), for identification of circulating microorganisms.

SUMMARY:
Rapid detection of microorganisms is a promising approach towards early administration of appropriate antibiotics for sepsis. This study aims to investigate the potential of a new NGS platform for the rapid diagnosis of circulating bacteria in blood.

DETAILED DESCRIPTION:
Early start of antimicrobials is the cornerstone of management of critically ill patients. The appropriate time window for this early intervention may vary greatly, but it is considered to be one to 3 hours from hospital admission. However, the choice of the antimicrobials for early intervention relies on empirical selection and may several times be inappropriate due to the emergence of antimicrobial resistance. The only way to overcome this difficulty is guidance through early microbial identification and antibiotic susceptibility testing (AST). However, blood cultures are positive in almost 20% of critically ill patients and AST may delay as much as 72 hours.

This means that another type of approach is warranted which will tackle the major limitation of standard-of-care (SoC) microbiology, namely, the need to incubate whole blood into flasks enriched with growth media which necessitates subculturing once a blood flask turns positive. It is evident that rapid identification of the pathogen followed by AST using whole blood without the need of blood culture can be a major advance in the diagnostic field.

The present study is based on previous analysis of ethylenediaminetetraacetic acid (EDTA) whole blood coming from patients with known bloodstream infection. Next generation sequencing (NGS) of bacterial DNA extracted from whole blood managed to identify the correct pathogen. This study is aiming at the validation of this NGS -based assay in a broader number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years.
* Both genders.
* Written informed consent provided by the patient or by one first-degree relative/spouse in case of patients unable to consent.
* Patients with high suspicion of infection with at least one sign of the quick SOFA score (i.e. one of mental confusion, more than 22 breaths per minute or systolic blood pressure less than 100mmHg).

Exclusion Criteria:

* Age below 18 years.
* Denial for written informed consent.
* Patients already receiving antibiotics.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet all inclusion criteria and who do not meet any exclusion criterion will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
The rate of matching between the results of Next Generation Sequencing and the Standard-of-Care culture for patients with sepsis. | 7 days
  This will be done by assessing the sensitivity, the specificity, the positive predictive value and the negative predictive value of Next Generation Sequencing and Standard-of-Care. For the analysis of this diagnostic performance, the results of the SoC cultures will be considered the "gold standard" for comparisons.

SECONDARY OUTCOMES:
Difference in time to identification of the bacterial pathogen between Next Generation Sequencing and the Standard-of-Care culture | 7 days
  The time from start of incubation until final identification will be recorded and compared between the two methods.
Difference in time to Antibiotic Susceptibility Testing between Next Generation Sequencing and the Standard-of-Care culture | 7 days
  The time from start of incubation until the Antibiotic Susceptibility Testing will be recorded and compared between the two methods.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD,PhD, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (4):
- Greece (4):
  - 4th Department of Internal Medicine,"Attikon" University Hospital, National and Kapodistrian University of Athens, Medical School, Chaïdári, Attica
  - 1st Department of Internal Medicine, General Hospital of Eleusis THRIASIO, Athens
  - 3rd University Department of Internal Medicine, General Hospital of Chest Diseases of Athens SOTIRIA, Athens
  - 3rd Department of Internal Medicine, General Hospital of Nikaia AGIOS PANTELEIMON, Nikaia

IPD SHARING:
Plan to Share IPD: No